CLINICAL TRIAL: NCT04091529
Title: A Prospective Study on Radiofrequency Ablation of Uterine Fibroids (Myolysis) Under Ultrasound and Endoscopic Guidance, in Single or Combined Approach
Brief Title: Tailored Radiofrequency Ablation of Uterine Myomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Evangelical Hospital (Other)
Responsible Party: Principal Investigator, Alessandro FASCIANI, MD - Principal Investigator, International Evangelical Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 295/2018
Record Dates: First submitted 2019-07-21; First posted 2019-09-16 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency myolysis of uterine fibroids (Experimental): 54 premenopausal participants with symptomatic uterine myomas
  Interventions: Device: RADIOFREQUENCY ABLATION OF UTERINE MYOMAS

INTERVENTIONS:
Device: RADIOFREQUENCY ABLATION OF UTERINE MYOMAS — The ablation device consisted of an radiofrequency (RF) energy generator (STARmed, RF generator VRS01) and an electric pump for the continuous cooling of the electrode tip. The RF generator to which the electrode (STARmed Gyeonggi-Do, Korea) is connected displays simultaneously the temperature of the electrode tip, the tissue impedance characteristics, the power and the ablation time. A 35 cm long 18Gauge internally cooled electrode with an exposed tip of 10 mm or a variable exposed tip was used
  Other Names: Radiofrequency myolysis (RFM); RF lesion generator for tissue ablation during surgical procedures. Sterile single-use RF coagulation monopolar electrode.

SUMMARY:
To perform the use of radiofrequency myolysis (RFM) for the treatment of intra-uterine fibroids through less invasive access by combining trans-vaginal ultrasound, hysteroscopy and laparoscopy

DETAILED DESCRIPTION:
Given that the RF ablation of solid tumors of the liver and other organs is successfully used as a usual approach, the investigators have decided to transfer this technology to an original treatment of uterine fibroids. The access to each individual fibroid was determined considering passage of the needle towards its centre through only compromised tissue and by the shortest possible route by combining trans-vaginal ultrasound, hysteroscopy and laparoscopy. To optimize radiofrequency myolysis, in fact, the investigators decided to improve the procedure by inserting three innovative elements: application of a virtual needle tracking system to follow the RF electrode during the ablation session, real-time monitoring of RF ablation by contrast-enhanced ultrasound and systematic biopsy of the lesions before electro-coagulation.

ELIGIBILITY:
"Inclusion Criteria":

* women who had symptomatic myomas with diameters ranging between 1.2 and 7.7 cm. - patients who had declined hysterectomy or laparoscopic myomectomy
* submucosal fibroids with intramural extension ≥50%
* intramural fibroids (FIGO G3 / G4 types)
* subserosal fibroids (FIGO G5 / G6 types)

"Exclusion Criteria":

* Women with intracavitary (FIGO G0 / G1 types) or subserosal-pedunculated fibroids / (FIGO G7 types)
* genital malignancy
* cervical dysplasias
* pelvic infection / adhesions
* severe systemic diseases
* pregnancy
* deeply infiltrating endometriosis
* patients who took gonadotropin-releasing hormone therapy or acetate ulipristal within 6 months

Ages: 30 Years to 62 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Myoma volumes after radiofrequency myolysis (RFM) | 12 months
  The outcomes evaluated after RFM were myoma volumes (cubic centimeters)
Myoma diameters after radiofrequency myolysis (RFM) | 12 months
  The outcomes evaluated after RFM were myoma diameters (centimeters)
Uterine Fibroid Symptom and Quality of Life (UFS-QOL) score after radiofrequency myolysis (RFM) | 12 months
  Uterine Fibroid Symptom and Quality of Life (UFS-QOL) questionnaire with scores ranging from 0 to 100, were higher QOL scores mean a better health-related QOL 1 and a 10-point scale used for each reported symptom.

SECONDARY OUTCOMES:
Surgical time of radiofrequency myolysis (RFM) | 12 months
  The surgical time (minutes) for each different type of surgical access
Surgical time of radiofrequency myolysis (RFM) assisted by new technologies | 12 months
  The reduction of surgical time (minutes) with the use of a virtual global positioning system (GPS) track system or a contrast-enhanced ultrasound during the ablation
Pre-intervention biopsy associated to radiofrequency myolysis (RFM) | 12 months
  The number of biopsies for treated fibroma

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro FASCIANI, Principal Investigator — International Evangelical Hospital
Locations (1):
- International Evangelical Hospital, Genoa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart EA, Lytle BL, Thomas L, Wegienka GR, Jacoby V, Diamond MP, Nicholson WK, Anchan RM, Venable S, Wallace K, Marsh EE, Maxwell GL, Borah BJ, Catherino WH, Myers ER. The Comparing Options for Management: PAtient-centered REsults for Uterine Fibroids (COMPARE-UF) registry: rationale and design. Am J Obstet Gynecol. 2018 Jul;219(1):95.e1-95.e10. doi: 10.1016/j.ajog.2018.05.004. Epub 2018 May 8. PMID 29750955
- [Background] Toub DB. A New Paradigm for Uterine Fibroid Treatment: Transcervical, Intrauterine Sonography-Guided Radiofrequency Ablation of Uterine Fibroids with the Sonata System. Curr Obstet Gynecol Rep. 2017;6(1):67-73. doi: 10.1007/s13669-017-0194-2. Epub 2017 Feb 15. PMID 28357157
- [Background] Yin G, Chen M, Yang S, Li J, Zhu T, Zhao X. Treatment of uterine myomas by radiofrequency thermal ablation: a 10-year retrospective cohort study. Reprod Sci. 2015 May;22(5):609-14. doi: 10.1177/1933719114556481. Epub 2014 Oct 29. PMID 25355802
- [Background] Lin L, Ma H, Wang J, Guan H, Yang M, Tong X, Zou Y. Quality of Life, Adverse Events, and Reintervention Outcomes after Laparoscopic Radiofrequency Ablation for Symptomatic Uterine Fibroids: A Meta-Analysis. J Minim Invasive Gynecol. 2019 Mar-Apr;26(3):409-416. doi: 10.1016/j.jmig.2018.09.772. Epub 2018 Sep 22. PMID 30253997
- [Result] Turtulici G, Orlandi D, Dedone G, Mauri G, Fasciani A, Sirito R, Silvestri E. Ultrasound-guided transvaginal radiofrequency ablation of uterine fibroids assisted by virtual needle tracking system: a preliminary study. Int J Hyperthermia. 2019 Jan 1;35(1):97-104. doi: 10.1080/02656736.2018.1479778. Epub 2018 Jul 17. PMID 30012030